CLINICAL TRIAL: NCT06733389
Title: Comparison of Peripheral Venous Pressure Variation, Pulse Pressure Variation and Pleth Variability Index in Predicting Fluid Responsiveness
Brief Title: Peripheral Venous Pressure Variation, Pulse Pressure Variation and Pleth Variability Index for Fluid Responsiveness
Status: Not yet recruiting | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Park InSun, Principal investigator, Seoul National University Bundang Hospital
Other Study IDs: B-2412-941-301
Record Dates: First submitted 2024-12-10; First posted 2024-12-13 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Pulse Pressure Variation; Stroke Volume Variation; Pleth Variability Index

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- peripheral waveform collection group: 1. Peripheral Venous Pressure Variation
  2. Pulse Pressure Variation
  3. Pleth Variability Index
  Interventions: Other: peripheral waveform collection

INTERVENTIONS:
Other: peripheral waveform collection — The peripheral venous pressure is collected by connecting a pressure transducer that is currently in use to the central venous line. In addition, pulse pressure variation and stroke volume variation that can be obtained from the arterial catheter. In addition, the pleth variability index is collected through the oxygen saturation monitoring. This extracts the medical records and bio-signal information of the subjects registered through the previously approved 'Establishment of a Bio-signal and Clinical Information Registry for the Development of Patient Monitoring Algorithms' (B-2202-738-401).

SUMMARY:
Pulse pressure variation (PPV) and pleth variability index (PVI) are widely used in clinical practice as indicators of the responsiveness to fluid therapy in patients receiving mechanical ventilation. PPV, which measures changes in arterial pressure, requires arterial puncture, which is invasive, and PVI, which detects subtle changes in oxygen saturation, requires an expensive, commercial monitoring equipment. In this study, we aimed to measure peripheral venous pressure variation using less invasive waveform variation in peripheral veins and to determine whether this indicator can be clinically used to predict the responsiveness to fluid therapy. In addition, the investigators aimed to confirm the superiority of the indicators by comparing them with the responsiveness to fluid therapy of the PPV and PVI.

DETAILED DESCRIPTION:
Pulse pressure variation (PPV) and pleth variability index (PVI) are widely used in clinical practice as indicators of the responsiveness to fluid therapy. The investigators aimed to measure peripheral venous pressure variation using less invasive waveform variation in peripheral veins and to determine whether this indicator can be clinically used to predict the responsiveness to fluid therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients voluntarily agreed and signed the written informed consent form before participating in the study
* Adults aged 19 years or older
* American Society of Anesthesiologists physical class (ASA) 1-3
* Patients scheduled for elective hepatectomy under general anesthesia
* Patients who require arterial pressure monitoring and additional peripheral venous access for routine anesthesia preparation
* Non-smokers with normal pulmonary function

Exclusion Criteria:

* Patients with abnormal findings on electrocardiogram before surgery
* Patients who cannot undergo peripheral venous puncture

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective hepatectomy under general anesthesia
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-12-28 (Estimated); Primary Completion 2025-11-28 (Estimated); Study Completion 2026-11-28 (Estimated)

PRIMARY OUTCOMES:
Fluid responsiveness | intraoperative period
  Cardiac output increases by more than 15% after 250 mL crystalloid injection during a fluid challenge

CONTACTS AND LOCATIONS:
Overall Officials: Insun Park, Principal Investigator — assistant professor
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyunggi-do, South Korea